CLINICAL TRIAL: NCT02206594
Title: Combined Cataract Surgery and Planned Descemetorhexis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Steve Koenig, Steven B. Koenig, MD, Medical College of Wisconsin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCW-EI-001
Record Dates: First submitted 2014-04-18; First posted 2014-08-01 (Estimated); Last update posted 2015-08-21 (Estimated); Status verified 2014-07

CONDITIONS: Fuchs' Corneal Dystrophy; Cataract
MeSH Terms: conditions — Fuchs' Endothelial Dystrophy; Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Descemetorhexis (Experimental)
  Interventions: Procedure: Descemetorhexis

INTERVENTIONS:
Procedure: Descemetorhexis

SUMMARY:
A pilot study designed to assess the feasibility of planned descemetorhexis for the treatment of Fuchs' corneal dystrophy.

ELIGIBILITY:
General Inclusion Criteria:

* Patient >18 years old
* Willing and able to provide informed consent

Ocular Inclusion Criteria (all ocular inclusion criteria apply only to the study eye):

* Fuchs' corneal dystrophy diagnosed
* Cataract present
* Best corrected visual acuity ≤ 20/40
* Candidate for current endothelial transplant procedure (DSAEK, DMEK)

General Exclusion Criteria:

* <18 years old
* Medically unstable patient
* Monocular patient
* Unwilling or unable to provide informed consent

Ocular Exclusion Criteria (all ocular exclusion criteria apply only to the study eye):

* Corneal dystrophy other than Fuchs'
* Central corneal scar or central opacity not related to Fuchs'
* Severe nonproliferative diabetic retinopathy or proliferative diabetic retinopathy
* History of prior vitreoretinal surgery
* Advanced or unstable glaucoma
* Known steroid responders with glaucoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2014-01; Primary Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Corneal clarity as assessed by slit lamp photography | Assessed up to 1 year following descemetorhexis

SECONDARY OUTCOMES:
Resolution of edema as assessed by slit lamp photography | Assessed up to 1 year following descemetorhexis

OTHER OUTCOMES:
Reconstitution of the endothelial cell layer as assessed by specular microscopy | Assessed up to 1 year following descemetorhexis

CONTACTS AND LOCATIONS:
Locations (1):
- The Medical College of Wisconsin, Milwaukee, Wisconsin, United States